CLINICAL TRIAL: NCT04315974
Title: Italian Registry In the Setting of AF Ablation With Rivaroxaban
Brief Title: Italian Registry In the Setting of AF Ablation With Rivaroxaban (IRIS)
Acronym: IRIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr Carlo Lavalle (Other)
Collaborators: Istituto Nazionale per le Ricerche Cardiovascolari (INRC) (Unknown)
Responsible Party: Sponsor-Investigator, Dr Carlo Lavalle, Medical Director at the Department of Cardiovascular, Respiratory, Nephrological, Anesthesiological and Geriatric Sciences., Azienda Policlinico Umberto I
Organization: Azienda Policlinico Umberto I (Other)
Other Study IDs: IRIS
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Atrial Fibrillation
Keywords: Catheter ablation; Rivaroxaban; Real-world clinical practice; Italian registry; Non-valvular Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; Catheter Ablation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nonvalvular atrial fibrillation patients (NVAF): Eligible patients comprise men and women aged 18 years or older with nonvalvular atrial fibrillation diagnosis undergoing ablation procedure.
  Interventions: Drug: Rivaroxaban; Procedure: Catheter ablation

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban therapy for at least 4 weeks.
Procedure: Catheter ablation — Radiofrequency catheter ablation or cryoballoon ablation.

SUMMARY:
The aim of IRIS study is to observe the safety and efficacy of Rivaroxaban in subjects undergoing catheter ablation for atrial fibrillation (AF) in real-world clinical practice.

The transcatheter ablation of AF is now considered an essential therapeutic strategy in the management of patients with this arrhythmia. In fact, it is known how fibrillating patients have a greater risk to develop thromboembolic phenomena; this risk can also increase during ablation (risk intrinsically with the procedure), therefore a careful anti-coagulant therapy is fundamental to avoid the formation of new thrombus and their dissemination through blood circulation.

The use of direct oral anti-coagulants (DOAC) in the fibrillating patient has been revealed a more safe and effective approach if compared with the standard therapy (direct vitamin K antagonists, VKA).

In the specific case of the Rivaroxaban, several experimental trials have shown how the uninterrupted administration of the drug before the ablation procedure is safe and valid. However, little information related to its use in the daily clinical assistance activity is still known and no real-life data are available for the Italian context.

Moreover, in Italy the uninterrupted strategy is not commonly used, and physicians often adopt the short interruption strategy.

Thus, the IRIS registry is aimed to collect new real-life data by collecting not only information regarding the effectiveness and safety of the drug, but also regarding the type of strategy (short interruption or uninterrupted strategy) used by the Italian centers participating to this study.

DETAILED DESCRIPTION:
IRIS study is an Italian, multicenter, prospective and non-interventional study aimed to observe the safety and efficacy of uninterrupted or shortly interrupted catheter ablation procedure with Rivaroxaban in nonvalvular atrial fibrillation (NVAF) patients in real-world clinical practice.

250 patients treated with rivaroxaban undergoing AF-ablation procedure are expected to be enrolled in two years. The patients can arrive already taking rivaroxaban or if they are naïve, the investigators will start the therapy and taking rivaroxaban for at least 4 weeks. The decision to prescribe rivaroxaban is under discretion of the treating physician, including the dose and duration of therapy. Also the decision on the ablation technique and energy used during the procedure (radiofrequency catheter ablation or Cryoballoon Ablation) is up to the investigators.

Because this study is intended to assess the use of rivaroxaban in routine real-world clinical practice, study protocol will not interfere with the clinical management of patients or with the prescribing behaviors of attending physicians.

IRIS study will include all consenting patients and collect data at the following time points:

* One inclusion/exclusion visit at the hospital (during hospitalization or outpatient visit);
* Ablation procedure in hospital;
* One-month follow-up visit.

Baseline Data

The Following information will be collected for each enrolled patient at the initial visit:

* Patient demographics (date of birth, gender, ethnic origin, height/weight)
* Previous therapies or interventions to treat AF, including cardioversion and ablation
* AF characteristics (paroxysmal or persistent)
* Cardiovascular risk factors, concomitant cardiovascular diseases and other diseases/conditions
* Concomitant medications
* Stroke and bleeding risk profiles based on CHA2DS2 (Congestive heart failure, Hypertension, Age, Diabetes Mellitus, Stroke) - VASc27 (Vascular disease, Age, Sex) score, and HAS (Hypertension, Abnormal renal and liver function, Stroke) - BLED28 (Bleeding, Labile International Normalized Ratio, Elderly, Drugs or alcohol) score.
* Data on the AF-related diagnostic assessment, including electrocardiographic assessment, blood biochemistry, echocardiography and other diagnostic procedures, if performed as part of routine care
* Inform consent signature

Ablation procedure

* Type of Ablation procedure
* Activated Clotting Time (ACT)
* Adverse Event (AE)/Serious Adverse Event (SAE)
* Major complication events

Follow-Up Data Follow-up data at 1 month will be collected for all patients.

The following information will be obtained by phone or during a visit to the center for each enrolled patient:

* Any bleedings event described in the study protocol;
* Major complications described in the study protocol;
* Adherence to Non-VKA Oral Anticoagulant (NOACs) therapy,
* Concomitant medications;
* Concomitant procedures;
* AE/SAE.

ELIGIBILITY:
Inclusion Criteria:

* Suitable for anticoagulant therapy and catheter ablation;
* Scheduled for Non Valvular Atrial Fibrillation (NVAF) catheter ablation;
* Paroxysmal or persistent NVAF;
* Patient naïve or in therapy with Rivaroxaban;
* Written informed consent.

Exclusion Criteria:

* Patients who do not agree with study inclusion;
* Impossible to Non-VKA Oral Anticoagulant (NOAC);
* Moderate to severe hepatic impairment;
* Pregnancy or lactation;
* Creatinine Clearance (CrCl) < 15 ml/min.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients comprise men and women aged 18 years or older with nonvalvular atrial fibrillation (AF) diagnosis undergoing ablation procedure.
  250 patients treated with rivaroxaban undergoing AF-ablation procedure will be enrolled. The patients can arrive already taking rivaroxaban or, if they are naïve, the investigators will start the therapy and taking rivaroxaban for at least 4 weeks. The decision to prescribe rivaroxaban is under discretion of the treating physician, including the dose and duration of therapy.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of thromboembolic and bleeding events. | 30 ± 5 days after the catheter ablation procedure.
  Thromboembolic events:
  * Ischemic stroke;
  * Vascular death.
  Major bleeding events:
  * Fatal bleeding;
  * Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome;
  * Bleeding causing a fall in hemoglobin level of 20 g L-1 or more, or leading to transfusion of two or more units of whole blood or red cells.
  Non-major clinically relevant bleeding events:
  overt bleeding not meeting the criteria for major bleeding but associated with medical intervention.

SECONDARY OUTCOMES:
Effectiveness endpoints | 30 days after the catheter ablation procedure.
  The secondary endpoint is the incidence of any of the below listed events within the first 30 days after the catheter ablation procedure:
  * Stroke;
  * Transient ischemic attack (TIA);
  * Myocardial infarction (MI);
  * Venous Thromboembolism (VTE).
Ablation procedure endpoints | 30 days after the catheter ablation procedure.
  The secondary endpoint is the incidence of any of the below listed events within the first 30 days after the catheter ablation procedure:
  * Death;
  * Tamponade;
  * Total femoral pseudoaneurysm;
  * Total artero-venous fistulae.

OTHER OUTCOMES:
Activated Clotting Time (ACT) | During the ablation procedure.
  ACT evaluation to assess procedural heparin dose requirement during the ablation procedure.
Study medication adherence | At baseline and after 30 days.
  The study medication adherence is evaluated counting pills from the blister at baseline and after 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Lavalle, Dr, Principal Investigator — Policlinico Umberto I
Locations (1):
- Azienda Ospedaliero-Universitaria Policlinico Umberto I - Dipartimento di Scienze Cardiovascolari, Respiratorie, Nefrologiche, Anestesiologiche e Geriatriche., Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
It has been planned to share all Individual Participant Data (IPD) that underlie results in a publication.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Lakkireddy D, Reddy YM, Di Biase L, Vallakati A, Mansour MC, Santangeli P, Gangireddy S, Swarup V, Chalhoub F, Atkins D, Bommana S, Verma A, Sanchez JE, Burkhardt JD, Barrett CD, Baheiry S, Ruskin J, Reddy V, Natale A. Feasibility and safety of uninterrupted rivaroxaban for periprocedural anticoagulation in patients undergoing radiofrequency ablation for atrial fibrillation: results from a multicenter prospective registry. J Am Coll Cardiol. 2014 Mar 18;63(10):982-8. doi: 10.1016/j.jacc.2013.11.039. Epub 2014 Jan 8. PMID 24412445
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2017 Oct;14(10):e275-e444. doi: 10.1016/j.hrthm.2017.05.012. Epub 2017 May 12. No abstract available. PMID 28506916
- [Background] Nairooz R, Sardar P, Pino M, Aronow WS, Sewani A, Mukherjee D, Paydak H, Maskoun W. Meta-analysis of risk of stroke and thrombo-embolism with rivaroxaban versus vitamin K antagonists in ablation and cardioversion of atrial fibrillation. Int J Cardiol. 2015;187:345-53. doi: 10.1016/j.ijcard.2015.03.323. Epub 2015 Mar 21. PMID 25839640
- [Background] Zhao Y, Yang Y, Tang X, Yu X, Zhang L, Xiao H. New oral anticoagulants compared to warfarin for perioperative anticoagulation in patients undergoing atrial fibrillation catheter ablation: a meta-analysis of continuous or interrupted new oral anticoagulants during ablation compared to interrupted or continuous warfarin. J Interv Card Electrophysiol. 2017 Apr;48(3):267-282. doi: 10.1007/s10840-016-0221-7. Epub 2017 Jan 12. PMID 28078536
- [Background] Romero J, Cerrud-Rodriguez RC, Diaz JC, Michaud GF, Taveras J, Alviz I, Grupposo V, Cerna L, Avendano R, Kumar S, Kirchhof P, Natale A, Di Biase L. Uninterrupted direct oral anticoagulants vs. uninterrupted vitamin K antagonists during catheter ablation of non-valvular atrial fibrillation: a systematic review and meta-analysis of randomized controlled trials. Europace. 2018 Oct 1;20(10):1612-1620. doi: 10.1093/europace/euy133. PMID 29982383
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Piccini JP, Stevens SR, Lokhnygina Y, Patel MR, Halperin JL, Singer DE, Hankey GJ, Hacke W, Becker RC, Nessel CC, Mahaffey KW, Fox KA, Califf RM, Breithardt G; ROCKET AF Steering Committee & Investigators. Outcomes after cardioversion and atrial fibrillation ablation in patients treated with rivaroxaban and warfarin in the ROCKET AF trial. J Am Coll Cardiol. 2013 May 14;61(19):1998-2006. doi: 10.1016/j.jacc.2013.02.025. Epub 2013 Mar 14. PMID 23500298
- [Background] Tao S, Otomo K, Ono Y, Osaka Y, Hirao T, Koura K, Manno T, Ueshima D, Shimizu S, Isobe M, Hirao K. Efficacy and safety of uninterrupted rivaroxaban taken preoperatively for radiofrequency catheter ablation of atrial fibrillation compared to uninterrupted warfarin. J Interv Card Electrophysiol. 2017 Mar;48(2):167-175. doi: 10.1007/s10840-016-0214-6. Epub 2016 Dec 9. PMID 27943112
- [Background] Dillier R, Ammar S, Hessling G, Kaess B, Pavaci H, Buiatti A, Semmler V, Kathan S, Hofmann M, Lennerz C, Kolb C, Reents T, Deisenhofer I. Safety of continuous periprocedural rivaroxaban for patients undergoing left atrial catheter ablation procedures. Circ Arrhythm Electrophysiol. 2014 Aug;7(4):576-82. doi: 10.1161/CIRCEP.114.001586. Epub 2014 Jun 26. PMID 24970293
- [Background] Cappato R, Marchlinski FE, Hohnloser SH, Naccarelli GV, Xiang J, Wilber DJ, Ma CS, Hess S, Wells DS, Juang G, Vijgen J, Hugl BJ, Balasubramaniam R, De Chillou C, Davies DW, Fields LE, Natale A; VENTURE-AF Investigators. Uninterrupted rivaroxaban vs. uninterrupted vitamin K antagonists for catheter ablation in non-valvular atrial fibrillation. Eur Heart J. 2015 Jul 21;36(28):1805-11. doi: 10.1093/eurheartj/ehv177. Epub 2015 May 14. PMID 25975659
- [Background] Aryal MR, Ukaigwe A, Pandit A, Karmacharya P, Pradhan R, Mainali NR, Pathak R, Jalota L, Bhandari Y, Donato A. Meta-analysis of efficacy and safety of rivaroxaban compared with warfarin or dabigatran in patients undergoing catheter ablation for atrial fibrillation. Am J Cardiol. 2014 Aug 15;114(4):577-82. doi: 10.1016/j.amjcard.2014.05.038. Epub 2014 Jun 6. PMID 24998087
- [Background] Li W, Gao C, Li M, Wang X, Qi D, Zhang Y, Hao P, Liu J, Zhu L. Safety and efficacy of rivaroxaban versus warfarin in patients undergoing catheter ablation of atrial fibrillation: a meta-analysis of observational studies. Discov Med. 2015 Mar;19(104):193-201. PMID 25828523
- [Background] Phan K, Wang N, Pison L, Kumar N, Hitos K, Thomas SP. Rivaroxaban versus warfarin or dabigatran in patients undergoing catheter ablation for atrial fibrillation: A meta-analysis. Int J Cardiol. 2015 Apr 15;185:209-13. doi: 10.1016/j.ijcard.2015.03.102. Epub 2015 Mar 10. No abstract available. PMID 25797679
- [Background] Camm AJ, Amarenco P, Haas S, Hess S, Kirchhof P, Kuhls S, van Eickels M, Turpie AG; XANTUS Investigators. XANTUS: a real-world, prospective, observational study of patients treated with rivaroxaban for stroke prevention in atrial fibrillation. Eur Heart J. 2016 Apr 7;37(14):1145-53. doi: 10.1093/eurheartj/ehv466. Epub 2015 Sep 1. PMID 26330425
- [Background] Hecker J, Marten S, Keller L, Helmert S, Michalski F, Werth S, Sahin K, Tittl L, Beyer-Westendorf J. Effectiveness and safety of rivaroxaban therapy in daily-care patients with atrial fibrillation. Results from the Dresden NOAC Registry. Thromb Haemost. 2016 May 2;115(5):939-49. doi: 10.1160/TH15-10-0840. Epub 2016 Jan 21. PMID 26791999
- [Background] Tamayo S, Frank Peacock W, Patel M, Sicignano N, Hopf KP, Fields LE, Sarich T, Wu S, Yannicelli D, Yuan Z. Characterizing major bleeding in patients with nonvalvular atrial fibrillation: a pharmacovigilance study of 27 467 patients taking rivaroxaban. Clin Cardiol. 2015 Feb;38(2):63-8. doi: 10.1002/clc.22373. Epub 2015 Jan 14. PMID 25588595
- [Background] Coleman CI, Antz M, Bowrin K, Evers T, Simard EP, Bonnemeier H, Cappato R. Real-world evidence of stroke prevention in patients with nonvalvular atrial fibrillation in the United States: the REVISIT-US study. Curr Med Res Opin. 2016 Dec;32(12):2047-2053. doi: 10.1080/03007995.2016.1237937. Epub 2016 Sep 20. PMID 27633045
- [Background] Camm AJ, Turpie AGG, Hess S, Amarenco P, Lambelet M, Haas S, van Eickels M, Kirchhof P; XANTUS Investigators. Outcomes after catheter ablation and cardioversion in patients with non-valvular atrial fibrillation: results from the prospective, observational XANTUS study. Europace. 2018 Jun 1;20(6):e87-e95. doi: 10.1093/europace/eux127. PMID 29016755
- [Background] Sugrue A, Siontis KC, Piccini JP, Noseworthy PA. Periprocedural Anticoagulation Management for Atrial Fibrillation Ablation: Current Knowledge and Future Directions. Curr Treat Options Cardiovasc Med. 2018 Jan 25;20(1):3. doi: 10.1007/s11936-018-0600-8. PMID 29368193
- [Background] Sawhney V, Shaukat M, Volkova E, Jones N, Providencia R, Honarbakhsh S, Dhillon G, Chow A, Lowe M, Lambiase PD, Dhinoja M, Sporton S, Earley MJ, Schilling RJ, Hunter RJ. Catheter ablation for atrial fibrillation on uninterrupted direct oral anticoagulants: A safe approach. Pacing Clin Electrophysiol. 2018 May 16. doi: 10.1111/pace.13370. Online ahead of print. PMID 29768672
- [Background] Yoshimura A, Iriki Y, Ichiki H, Oketani N, Okui H, Maenosono R, Namino F, Miyata M, Ohishi M. Evaluation of safety and efficacy of periprocedural use of rivaroxaban and apixaban in catheter ablation for atrial fibrillation. J Cardiol. 2017 Jan;69(1):228-235. doi: 10.1016/j.jjcc.2016.03.014. Epub 2016 Apr 27. PMID 27131792
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Cappato R, Calkins H, Chen SA, Davies W, Iesaka Y, Kalman J, Kim YH, Klein G, Natale A, Packer D, Skanes A, Ambrogi F, Biganzoli E. Updated worldwide survey on the methods, efficacy, and safety of catheter ablation for human atrial fibrillation. Circ Arrhythm Electrophysiol. 2010 Feb;3(1):32-8. doi: 10.1161/CIRCEP.109.859116. Epub 2009 Dec 7. PMID 19995881
- [Background] Lip GY, Nieuwlaat R, Pisters R, Lane DA, Crijns HJ. Refining clinical risk stratification for predicting stroke and thromboembolism in atrial fibrillation using a novel risk factor-based approach: the euro heart survey on atrial fibrillation. Chest. 2010 Feb;137(2):263-72. doi: 10.1378/chest.09-1584. Epub 2009 Sep 17. PMID 19762550
- [Background] Pisters R, Lane DA, Nieuwlaat R, de Vos CB, Crijns HJ, Lip GY. A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest. 2010 Nov;138(5):1093-100. doi: 10.1378/chest.10-0134. Epub 2010 Mar 18. PMID 20299623
- [Background] Fleiss JL, Levin B, Paik MC. Statistical methods for rates and proportions (3rd edn). Wiley, New Jersey, 2003.
- [Background] Newcombe RG. Two-sided confidence intervals for the single proportion: comparison of seven methods. Stat Med. 1998 Apr 30;17(8):857-72. doi: 10.1002/(sici)1097-0258(19980430)17:83.0.co;2-e. PMID 9595616
- [Background] Velu S, Pathiraja J, Barr C, Forsey P, Lapper A, Kidd G, Arya A, Petkar S. A wide range of catheter ablations can be safely performed without interrupting novel oral anticoagulants (NOAC's). EP Europace, Volume 19, Issue suppl_3, 1 June 2017, Page iii298